CLINICAL TRIAL: NCT04879992
Title: Rifabutin-containing Triple Therapy for Rescue Treatment of Helicobacter Pylori: A Randomized Clinical Trial
Brief Title: Rifabutin-containing Triple Therapy for Treatment of Helicobacter Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjcjn20210506
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori Therapy
MeSH Terms: interventions — Esomeprazole; Tetracycline; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetracycline Bismuth Quadruple Therapy (Active Comparator): Esomeprazole 20mg bid, Bismuth Potassium Citrate 300mg bid, Tetracycline 500mg qid, Metronidazole 400mg qid
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Tetracycline,Metronidazole
- rifabutin triple therapy (Experimental): Esomeprazole 20mg bid, amoxicillin 1000mg bid, rifabutin 150mg bid
  Interventions: Drug: Esomeprazole; Drug: amoxicillin rifabutin

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
  Arms: Tetracycline Bismuth Quadruple Therapy
Drug: Tetracycline,Metronidazole — Antibiotics for H. pylori eradication
  Arms: Tetracycline Bismuth Quadruple Therapy
Drug: amoxicillin rifabutin — Antibiotics for H. pylori eradication
  Arms: rifabutin triple therapy

SUMMARY:
Rifabutin has good chemical stability and low drug resistance rate in acidic gastric environment. Therefore, it is often used in combination with amoxicillin proton pump inhibitor for the rescue treatment of Helicobacter pylori. The purpose of this study was to evaluate the efficacy and safety of rifabutin-containing triple therapy versus classical bismuth-containing quadruple therapy as rescue therapy for the eradication of refractory Helicobacter pylori

ELIGIBILITY:
Inclusion Criteria:

* ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection and with previous treatment experience

Exclusion Criteria:

* Less than 18 years old
* With previous gastric surgery
* Previous history of tuberculosis
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was

SECONDARY OUTCOMES:
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Guo Y, Huang Y, Ding Z, Wang J, Liang X, Xu P, Han Y, Lu H. Rifabutin-Containing Triple Therapy Versus Bismuth Quadruple Therapy for Helicobacter pylori Rescue Treatment: A Multicenter, Randomized Controlled Trial. J Infect Dis. 2023 Aug 31;228(5):511-518. doi: 10.1093/infdis/jiad114. PMID 37079894